CLINICAL TRIAL: NCT01451944
Title: Effect of Home Health Nurse Case Management on Asthma Morbidity
Brief Title: Effect of Home Health Case Management on Asthma Morbidity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no one enrolled
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Judith A Theriot, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11.0320
Record Dates: First submitted 2011-10-04; First posted 2011-10-14 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Asthma; Childhood Asthma
Keywords: Asthma; Home Health Nursing; Patient education
MeSH Terms: conditions — Asthma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- asthma education and case management (Experimental): asthma education and case management
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — home asthma case management and education

SUMMARY:
The objective of our program is to evaluate the effect of home health nurse intervention and education on hospital admissions, ER utilization and asthma control of Passport asthma patients. The investigators hypothesize that case management and in home education by nurses will decrease hospitalizations and ER asthma visits and improves disease control in our population.

Our clinic population consists of primarily inner-city, low income, medicaid recipients. This population suffers from severe asthma much more than the typical pediatric population. Asthma remains the most frequent cause of hospital admission for our patient population. Home health nurse asthma education and home visits have been reported to reduce asthma triggers in the home and improve asthma control. The unique partnership between the pediatrician and the home health nurse will give us a better understanding of the health needs for this population, will improve quality of care and deliver more cost effective care.

DETAILED DESCRIPTION:
Asthma patients age 3-17 enrolled in our clinic who have been seen in the ER, hospital or clinic for an asthma exacerbation will be invited to participate. Once enrolled they will have a home health nurse visit their home and provide medical assessment, asthma education and determine if the patients has all needed medications available. They enrolled patient will receive another home visit at 1, 4, and 12 months after enrollment. The medical record will be reviewed and ER visits and hospitalizations recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3-17 years with asthma who attend our clinic who present with an asthma exacerbation to the clinic, ER or hospital.

Exclusion Criteria:

* Patients with airway anomalies or tracheostomy

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Decreased asthma hospitalization rates | 1 year
  patients will be followed for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Theriot, MD, Principal Investigator — University of Louisville
Locations (1):
- Children and Youth Project, Louisville, Kentucky, United States